CLINICAL TRIAL: NCT04188535
Title: RELAY: Repeated Magnetic Resonance Imaging Examinations to Analyze and Assess Your Cancer: A Prospective Study on the Use of Serial Magnetic Resonance Imaging in the Assessment of Changes During Treatment With Radiation Therapy
Brief Title: Serial MRI Scans During Radiation Therapy
Acronym: RELAY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jonathan Leeman, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 19-573
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Esophageal Cancer; Radiotherapy; Magnetic Resonance Imaging; MRI; Prostate Cancer; Vulvar Cancer; Pediatric Glioblastoma Multiforme
Keywords: Glioblastoma; Esophageal Cancer; Radiotherapy; Magnetic Resonance Imaging; MRI; Prostate Cancer; Vulvar Cancer; Pediatric Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma; Esophageal Neoplasms; Prostatic Neoplasms; Vulvar Neoplasms; Astrocytoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (8):
- Esophageal Cohort (Experimental): The research study procedures include:
  * Screening for eligibility
  * Three MRI scans (prior to start of standard cancer treatment, in the middle, and at the end of radiation treatment). Imaging with MRI will be performed as per disease site standards.
  Interventions: Diagnostic Test: MRI IMAGING
- Glioblastoma Cohort (Experimental): The research study procedures include:
  * Screening for eligibility
  * Three MRI scans prior to start of standard cancer treatment, in the middle, and at the end of radiation treatment). Imaging with MRI will be performed as per disease site standards.
  Interventions: Diagnostic Test: MRI IMAGING
- Glioblastoma Expansion Cohort Serial MR Imaging Registry (Experimental): The research study procedures include:
  * Screening for eligibility
  * Three MRI scans prior to start of standard cancer treatment, in the middle, and at the end of radiation treatment). Imaging with MRI will be performed as per disease site standards.
  Interventions: Diagnostic Test: MRI IMAGING
- Prostate Cancer Cohort (Experimental): The research study procedures include:
  * Screening for eligibility
  * Three MRI scans prior to start of androgen deprivation therapy, prior to the start of radiation treatment, and after radiation treatment). Imaging with MRI will be performed as per disease site standards.
  * Genomic testing of biopsy sample
  Interventions: Diagnostic Test: MRI IMAGING
- Prostate Cancer Expansion Cohort Serial MR Imaging Registry (Experimental): The research study procedures include:
  * Screening for eligibility
  * Three MRI scans prior to start of androgen deprivation therapy, prior to the start of radiation treatment, and after radiation treatment). Imaging with MRI will be performed as per disease site standards.
  * Genomic testing of biopsy sample
  Interventions: Diagnostic Test: MRI IMAGING
- Vulvar Cancer Cohort (Experimental): The research study procedures include:
  * Screening for eligibility
  * Three MRI scans prior to start of standard cancer treatment, in the middle, and at the end of radiation treatment). Imaging with MRI will be performed as per disease site standards.
  Interventions: Diagnostic Test: MRI IMAGING
- Pediatric Glioma Cohort (Experimental): The research study procedures include:
  * Screening for eligibility
  * Three MRI scans prior to start of standard cancer treatment, in the middle, and at the end of radiation treatment). Imaging with MRI will be performed as per disease site standards.
  Interventions: Diagnostic Test: MRI IMAGING
- Sarcoma Cohort (Experimental): The research study procedures include: • Screening for eligibility • Three MRI scans prior to start of standard cancer treatment, in the middle, and at the end of radiation treatment). Imaging with MRI will be performed as per disease site standards.
  Interventions: Diagnostic Test: MRI IMAGING

INTERVENTIONS:
Diagnostic Test: MRI IMAGING — Imaging with MRI will be performed as per disease site standards.

SUMMARY:
This is a phase 1 study to determine the feasibility and utility of using serial magnetic resonance imaging (MRI) to assess treatment response during and after radiation therapy (standard of care cancer treatment) for participants with advanced esophageal cancer, glioblastoma, prostate cancer, vulvar cancer or pediatric glioma.

The research study procedures include three MRI scans (one before, one during, and one after standard of care cancer radiation therapy) for participants with advanced esophageal cancer, glioblastoma, prostate cancer, vulvar cancer or pediatric glioma.

The research study procedures include:

* Screening for eligibility
* Three MRI scans

DETAILED DESCRIPTION:
This is a phase 1, non-randomized, open-label study evaluating feasibility of serial MRI, with an option for an expansion cohort. The optional expansion cohort is a prospective imaging registry evaluating imaging biomarkers as predictors of disease control with standard of care treatment.

This research study is a feasibility study, meaning that it is the first time that investigators at this institution are examining the process of getting multiple MRIs during radiation treatment.

The U.S. Food and Drug Administration (FDA) has cleared this MRI scanner for use.

Participants who fulfill eligibility criteria will be entered into the trial.

The research study procedures include screening for eligibility, and three MRI scans. MRI imaging will be performed as per disease site standards.

A total of 149 participants will be enrolled in this trial:

* 13 participants in the esophageal cancer cohort
* 10 participants in the initial glioblastoma cohort and 36 participants in the image registry expansion cohort
* 10 participants in the prostate cancer cohort and 50 participants in the image registry expansion cohort
* 10 participants in the vulvar cancer cohort
* 10 participants in the pediatric glioma cohort
* 10 participants in the sarcoma cohort

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed malignancy requiring radiation therapy.
* Age: 18 years or older except where otherwise specified in subprotocol.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Ability to understand and the willingness to sign a written informed consent document.
* Any further criteria listed in the specific disease site subprotocol.
* (Esophageal cohort) Patients must be considered appropriate candidates for neoadjuvant chemoradiation therapy followed by esophagectomy. Patients must have an endoscopic ultrasound done or scheduled to be done at the baseline visit.
* (Glioblastoma cohort) Patients with a histologically confirmed newly diagnosed intracranial glioblastoma or gliosarcoma who will be undergoing radiation therapy as part of clinical care.
* (Prostate cohort) Patients with localized prostate cancer who are planning to receive androgen deprivation therapy and definitive radiation therapy.
* (Vulvar cohort) Patients with biopsy-proven locally advanced vulvar cancer for which definitive radiotherapy is planned.
* (Pediatric glioma cohort) Patients age 18 or under (patients 18-30 years old are also eligible if the physician determines that based on genetics, the tumor biology is consistent with pediatric high grade glioma). Patients with a histologically confirmed newly diagnosed high-grade glioma (WHO grade III or IV) who will be undergoing radiation therapy as part of clinical care. Patients with DIPG are only eligible if biopsy-confirmed high grade DIPG is present. Ability to understand and/or willingness of their parent or legally authorized representative to sign a written informed consent document.

Exclusion Criteria:

* Disease-specific exclusion criteria will be specified in a subprotocol.
* For MRI involving contrast, history of allergic reactions attributed to gadolinium-based IV contrast. If patient will not receive contrast, this is not applicable and kidney function will not affect eligibility.
* Inability to undergo magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of acquiring serial MRI scans on an MRI simulator during treatment with radiation therapy | 1 year
  90% lower confidence limit (LCL) on the true feasibility rate. Feasibility is defined as successfully enrolling patients, acquiring MRI data at all timepoints, identifying the target on MRI data obtained at all timepoints, and processing MRI data at all timepoints to yield pre-specified MRI-derived measurements.
Ability to measure disease control (for imaging registry expansion cohort) | 2 years
  Validating a previously developed predictive model to identify the most likely area of recurrence using MRI-based features.

SECONDARY OUTCOMES:
Dosimetric change | 1 year
  For subprotocols studying the adaptive treatment, the secondary objective is dosimetric change in the in silico adaptive radiation therapy plans, without delivering adaptive plans in Phase I.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leeman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu